CLINICAL TRIAL: NCT01503762
Title: Mirror Therapy in Patients With Hand Orthopedic Disorders
Brief Title: Mirror Therapy and Hand Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamid Reza Rostami, Ms.C. Lecturer of Occupational Therapy Department, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pht-9006
Record Dates: First submitted 2011-12-04; First posted 2012-01-04 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Hand Fractures
Keywords: Hand Flexor tendon Injuries; hand Extensor Tendon Injuries; Hand Joint Dislocations and subluxation
MeSH Terms: conditions — Joint Dislocations | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirror Therapy Group (Experimental): Mirror Therapy Group
  Interventions: Other: Mirror therapy
- Control Group (Sham Comparator): Control Group receive classical rehabilitation techniques including splinting, tendon gliding, ...
  Interventions: Other: Classical rehabilitation techniques

INTERVENTIONS:
Other: Mirror therapy — mirror therapy
  Arms: Mirror Therapy Group
Other: Classical rehabilitation techniques — splinting, tendon gliding, active range of motion, activities of daliy living
  Arms: Control Group

SUMMARY:
Objective: The purpose of this study is to determine effects of mirror therapy in restoring hand function in patients with flexor lag following orthopedic injuries.

Methods: In a prospective randomized controlled trial, 22 patients with Flexor Lag will be measured. Intervention group will receive mirror therapy, 30-minute a day, 5 days a week for 3-week, as well, half an hour conventional rehabilitation after each mirror therapy session. Patients in the control group will receive the same treatment program, but instead of mirror, they will directly observe the affected hand. Outcome measures including Total Active Motion (TAM), and Disabilities of Arm, Shoulder and Hand (DASH) questionnaire will be administered before and after the treatment period and 3 weeks after the final treatment session.

ELIGIBILITY:
Inclusion Criteria:

* hand orthopedic Injuries
* more active range of motion than passive range of motion

Exclusion Criteria:

* crush injuries
* hand deformities
* not treated fractures and tendon ruptures
* complex regional pain syndrome
* psychiatric problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Total Active Motion | 6 Weeks
  Sum of Range of Motion in Metacarpophalangeal, Proximal Interphalangeal and Distal Interphalangeal Joints.

SECONDARY OUTCOMES:
Disabilities of the Shoulder, Arm, hand | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Reza Rostami, Principal Investigator — Ahvaz Jundishapur University of Medical Sciences
Locations (1):
- Musculoskeletal Rehabilitation Research Center, Ahvaz Jundishapur university of medical sciences, Ahvāz, Khouzestan, Iran

REFERENCES:
- [Derived] Rostami HR, Arefi A, Tabatabaei S. Effect of mirror therapy on hand function in patients with hand orthopaedic injuries: a randomized controlled trial. Disabil Rehabil. 2013 Sep;35(19):1647-51. doi: 10.3109/09638288.2012.751132. Epub 2013 Jan 22. PMID 23336124